CLINICAL TRIAL: NCT00521989
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate the Efficacy of CRx-102 in Subjects With Symptomatic Knee Osteoarthritis and Optional One-Year Extension
Brief Title: CRx-102 Osteoarthritis Multicenter Evaluation Trial
Acronym: COMET-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CRx-102-006 study results, negative
Sponsor: Zalicus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRx-102-006
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Results first posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; CRx-102; prednisolone; dipyridamole; CombinatoRx; WOMAC
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — dipyridamole, prednisolone drug combination; Prednisolone; Dipyridamole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- CRx-102 (2.7/90) (Experimental): 2.7 mg prednisolone plus 90 mg dipyridamole
  Subjects were dose twice daily through day 98. Prednisolone at 2.7 mg/d was administered as 1.8 mg at 8AM and 0.9 mg at 1PM. The dipyridamole dose was divided equally between the two time points, 8AM and 1PM
  Interventions: Drug: CRx-102 (2.7/90)
- CRx-102 (2.7/180) (Experimental): 2.7 mg prednisolone plus 180 mg dipyridamole
  Subjects were dose twice daily through day 98. Prednisolone at 2.7 mg/d was administered as 1.8 mg at 8AM and 0.9 mg at 1PM. The dipyridamole dose was divided equally between the two time points, 8AM and 1PM
  Interventions: Drug: CRx-102 (2.7/180)
- CRx-102 (2.7/360) (Experimental): 2.7 mg prednisolone plus 360 mg dipyridamole
  Subjects were dose twice daily through day 98. Prednisolone at 2.7 mg/d was administered as 1.8 mg at 8AM and 0.9 mg at 1PM. The dipyridamole dose was divided equally between the two time points, 8AM and 1PM
  Interventions: Drug: CRx-102 (2.7/90); Drug: CRx-102 (2.7/360)
- Prednisolone (Active Comparator): 2.7 mg prednisolone
  Subjects were dose twice daily through day 98. Prednisolone at 2.7 mg/d was administered as 1.8 mg at 8AM and 0.9 mg at 1PM.
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Placebo
  Subjects were dose twice daily through day 98.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRx-102 (2.7/90) — CRx-102 dose 1
  Other Names: 2.7 mg prednisolone plus 90 mg dipyridamole
  Arms: CRx-102 (2.7/360); CRx-102 (2.7/90)
Drug: Prednisolone — Prednisolone
  Other Names: 2.7 mg prednisolone
  Arms: Prednisolone
Drug: Placebo — Placebo
  Arms: Placebo
Drug: CRx-102 (2.7/180) — CRx-102 dose 2
  Other Names: Prednisolong 2.7 mg plus dipyridamole 180 mg
  Arms: CRx-102 (2.7/180)
Drug: CRx-102 (2.7/360) — CRx-102 dose 3
  Other Names: 2.7 mg prednisolone plus 360 mg dipyridamole
  Arms: CRx-102 (2.7/360)

SUMMARY:
CRx-102 is a synergistic combination drug candidate containing the cardiovascular drug dipyridamole and a very low dose of the glucocorticoid prednisolone. CRx-102 is believed to work through a novel mechanism of action in which dipyridamole selectively amplifies the anti-inflammatory and immunomodulatory activities of the glucocorticoid without replicating the dose-dependent adverse effects.

CRx-102 has been associated with clinical benefit in proof of concept studies in subjects with hand OA and RA. This is the first study to explore the efficacy of CRx-102 in knee OA. It is considered a dose-finding study and will also compare the potential benefits of CRx-102 treatment to both prednisolone administered alone and to placebo in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily give written informed consent
* Subject must be ≥ 40 years of age
* Knee pain for at least 6 months requiring NSAIDs or Coxibs for analgesia on the majority of days (≥ 15 days) during the preceding month
* WOMAC pain score when walking on a flat surface (question #1) between 30-80 mm at Screening with at least a 10 mm increase following NSAID or Coxib discontinuation during the Screening period
* Radiographic evidence of knee OA (Kellgren-Lawrence grade 2 or 3)
* Functional class I, II, or III according to the American Rheumatism Association
* Subject willing to take a multivitamin or the equivalent of at least 400 IU vitamin D and the equivalent of at least 1000 mg of elemental calcium daily

Exclusion Criteria:

* Predominant patellofemoral disease or clinically significant trauma to index knee
* History of clinically significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, osteoporotic and/or other major disease
* History of malignancy within the past 10 years (except for excised or treated basal cell or fewer than 3 squamous cell skin carcinomas)
* History of lymphoma or chronic leukemia
* Moles or lesions that are currently undiagnosed, but are suspicious for malignancy
* Surgery within the previous 3 months (except for minor dental, and/or cosmetic procedures)
* History of drug or alcohol abuse (as defined by the Investigator)
* History of bleeding disorder
* History of GI bleeding within 5 years of Screening
* History of severe migraines or headaches
* History of glaucoma
* Visually compromising cataract
* Active diabetic retinopathy
* History of osteoporotic fracture
* History of opportunistic infection
* Serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to Screening
* Fever or symptomatic viral or bacterial infection within 2 weeks prior to Screening
* Positive for hepatitis C (HCV) antibody
* Positive for hepatitis B surface antigen (HBsAg)
* Known positive history for human immunodeficiency virus (HIV) antibody
* Surgery on the index knee within 1 year of Screening
* History of hypersensitivity to steroids or dipyridamole
* Treatment with oral, intramuscular, or intravenous glucocorticoids within 6 weeks prior to Screening; intra-articular glucocorticoids within 10 weeks prior to Screening; inhaled glucocorticoid is permitted
* Treatment with injectable hyaluronic acid within 3 months of Screening
* Treatment with another investigational drug, investigational device, or approved therapy for investigational use within 30 days prior to Screening
* Treatment with NSAIDs (oral or topical), Coxibs or topical capsaicin
* Treatment with anticoagulants including: dipyridamole, warfarin, clopidogrel, ticlopidine, or ASA > 81 mg per day
* Treatment with any concomitant medications that have not been at a stable dose for at least 28 days prior to Screening
* Treatment for osteoporosis such as bisphosphonates (e.g., Fosamax®, Actonel®), or teriparatide (e.g., Forteo®), or calcitonin (e.g., Miacalcin, Calcimar) must be at stable dosages for at least 3 months prior to Screening
* ALT or AST laboratory values >1.5 X the ULN
* HgbA1c value of >7.0%
* Current enrollment in any other study with investigational drug or device
* Female subject who is pregnant or lactating
* Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for follow-up visits on schedule
* Other unspecified reasons that, in the opinion of the Investigator or sponsor make the subject unsuitable for enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Lee, PhD, Study Director — Zalicus
Locations (58):
- United States (57):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tuscon, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Rancho Mirage, California
  - Upland, California
  - Westlake Village, California
  - DeLand, Florida
  - Jupiter, Florida
  - Kissimee, Florida
  - Largo, Florida
  - Longwood, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Paducah, Kentucky
  - Covington, Louisiana
  - Towson, Maryland
  - Brockton, Massachusetts
  - Haverhill, Massachusetts
  - Peabody, Massachusetts
  - Worcester, Massachusetts
  - Bingham Farms, Michigan
  - Missoula, Montana
  - Reno, Nevada
  - Haddon Heights, New Jersey
  - Voorhees Township, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Plainview, New York
  - Rochester, New York
  - Hickory, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Mayfield Village, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Duncansville, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Cumberland, Rhode Island
  - Warwick, Rhode Island
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Sandy City, Utah
  - Roanoke, Virginia
  - Virginia Beach, Virginia
  - Tacoma, Washington
- Kitchener, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- CRx-102 (2.7/90 mg): CRx-102 (Prednisolone 2.7 mg + Dipyridamole 90 mg)
  prednisolone + dipyridamole: CRx-102 (Dose 1), CRx-102 (Dose 2), CRx-102 (Dose 3)
- CRx-102 (2.7/180 mg): CRx-102 Dose 2 (2.7 mg prednisolone + 180 mg dipyridamole)
  prednisolone + dipyridamole: CRx-102 (Dose 1), CRx-102 (Dose 2), CRx-102 (Dose 3)
- CRx-102 (2.7/360 mg): CRx-102 Dose 3 (2.7 mg prednisolone + 360 mg dipyridamole)
  prednisolone + dipyridamole: CRx-102 (Dose 1), CRx-102 (Dose 2), CRx-102 (Dose 3)
- Prednisolone: Prednisolone 2.7 mg
  Prednisolone: Prednisolone
Period: Overall Study
Arm/Group | CRx-102 (2.7/90 mg) | CRx-102 (2.7/180 mg) | CRx-102 (2.7/360 mg) | Prednisolone | Placebo
Started | 56 | 54 | 57 | 54 | 58
Completed | 36 | 37 | 41 | 42 | 35
Not Completed | 20 | 17 | 16 | 12 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRx-102 (2.7/90 mg) | CRx-102 (2.7/180 mg) | CRx-102 (2.7/360 mg) | Prednisolone | Placebo | Total
Number analyzed (Participants) | 56 | 54 | 57 | 54 | 58 | 279
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.35) | 59.4 (10.02) | 57.7 (9.03) | 60.2 (8.65) | 57.9 (7.46) | 59.3 (8.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 38 | 30 | 37 | 175
  Male | 19 | 21 | 19 | 24 | 21 | 104

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 98 Using the WOMAC Pain Question #1
Description: The WOMAC Index is a validated, 24-question self-administered assessment of three dimensions of pain, stiffness, and physical function for subjects with knee or hip OA. The WOMAC pain question #1 asks subjects to "think about the pain you felt in your (study joint) caused by your arthritis during the last 48 hours when walking on a flat surface." This is a visual analog scale (VAS) where the subject indicates pain severity by making a mark through a 100 mm horizontal line with "No Pain" on the left (0 mm) and "Extreme Pain" on the right (100 mm). The distance between the left end of the scale and the subject's mark is measured in millimeters. Lower values represent a better outcome.
Time Frame: Baseline to Day 98
Population: ITT population
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | CRx-102 (2.7/90 mg) | CRx-102 (2.7/180 mg) | CRx-102 (2.7/360 mg) | Prednisolone | Placebo
Number analyzed (Participants) | 56 | 54 | 57 | 54 | 58
millimeters | -32.4 (27.07) | -33.2 (32.02) | -37.3 (33.07) | -40.4 (30.04) | -34.6 (27.11)

2. Secondary Outcome: To Assess the Efficacy of the CRx-102 Compared to Placebo on the Change From Baseline to Day 98 Using the Full WOMAC Pain, Stiffness, Physical Function Parameters, and Patient Global Assessment VAS.
Time Frame: Day 98
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Prednisolone: Prednisolone 2.7 mg
- CRx-102 (2.7/90 mg): CRx-102 dose 1 (2.7 mg prednisolone + 90 mg dipyridamole)
- CRx-102 (2.7/180 mg): CRx-102 dose 2 (2.7 mg prednisolone + 180 mg dipyridamole)
- CRx-102 (2.7/360 mg): CRx-102 dose 3 (2.7 mg prednisolone + 360 mg dipyridamole)
Arm/Group | Placebo | Prednisolone | CRx-102 (2.7/90 mg) | CRx-102 (2.7/180 mg) | CRx-102 (2.7/360 mg)
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/54 | 2/56 | 1/54 | 1/57
Other Adverse Events (participants affected / at risk) | 19/58 | 26/54 | 29/56 | 29/54 | 40/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Prednisolone (N=54) | CRx-102 (2.7/90 mg) (N=56) | CRx-102 (2.7/180 mg) (N=54) | CRx-102 (2.7/360 mg) (N=57)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=58) | Prednisolone (N=54) | CRx-102 (2.7/90 mg) (N=56) | CRx-102 (2.7/180 mg) (N=54) | CRx-102 (2.7/360 mg) (N=57)
Headache (Nervous system disorders) | 10 | 14 | 16 | 17 | 28
Diarrhea (Gastrointestinal disorders) | 3 | 4 | 2 | 4 | 3
Nausea (Gastrointestinal disorders) | 4 | 3 | 0 | 4 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 4 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 2 | 1
Fatigue (General disorders) | 0 | 1 | 3 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days